CLINICAL TRIAL: NCT01204034
Title: Open-label, Prospective Exploratory Study to Assess the Effects of Formoterol and Beclometasone Dipropionate Combination Therapy on Central and Peripheral Airway Dimensions in COPD Patients
Brief Title: Study to Assess the Effect of Formoterol and Beclomethasone Dipropionate in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Wilfried De Backer, MD PhD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PML-DOC-1003; 2010-019864-36 (EudraCT Number)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Formoterol; Beclomethasone Dipropionate; Computational Fluid Dynamics; Functional Imaging; Central and Peripheral Airways; BODE index; COPD Assessment Test (CAT); Borg CR10 scale
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inuvair (Other)
  Interventions: Drug: Inuvair

INTERVENTIONS:
Drug: Inuvair — 6 µg formoterol and 100 µg beclometasone dipropionate combination spray pMDI aerosol

SUMMARY:
The objective of this study is to evaluate the effect of the combination of formoterol and beclometasone dipropionate on central and peripheral airway dimensions in COPD patients using Computational Fluid Dynamics (CFD). Further more, the effect of this combination therapy on lung function (spirometry, body plethysmography), the BODE index, COPD assessment test (CAT) and Borg CR10 scale will be assessed and the safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented COPD based on the following criteria:

Smoking history of at least 10 pack-years Decreased Tiffeneau index: FEV1/FVC < 0.70

* Male or female patients aged ≥ 40 years
* Patients should be treated according to the 'Global initiative for chronic Obstructive Lung Disease' (GOLD) guidelines
* Patients who present
* Moderate COPD with an FEV1 between 50 and 80% of predicted GOLD 2)
* Severe COPD with an FEV1 between 30 and 50% of predicted (GOLD 3)
* Very severe COPD with an FEV1 lower than 30% of predicted (GOLD 4)
* Patients will be maintained on stable respiratory medications for 6 weeks prior to screening
* Patients with a co-operative attitude and ability to be trained to correctly use the pMDI
* Written informed consent obtained

Exclusion Criteria:

* Pregnant or lactating females or females at risk of pregnancy
* Unstable patients who developed an exacerbation during the last 4 weeks
* Inability to carry out pulmonary function testing
* Diagnosis of asthma as defined by the current 'Global Initiative for Asthma' (GINA) guidelines
* Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
* Patients with a QTc interval (Bazett's formula) at the screening visit electrocardiogram (ECG) test >450 msec
* Cancer or any other chronic disease with poor prognosis and /or affecting patient status
* History of alcohol or drug abuse
* Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients
* Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
* Patients who received any investigational new drug within the last 4 weeks prior to the screening visit
* Patients treated with any non-permitted concomitant medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Peripheral airway resistance (from 4th bifurcation on) for the segmented airways | at baseline and after 6 months of treatment
Total airway volume for the segmented airways | at baseline and after 6 months of treatment
Peripheral airway volume (from the 4th bifurcation on) for the segmented airways | at baseline and after 6 months of treatment
Relative compliance for each lobe | at baseline and after 6 months of treatment
Density of the lung parenchyma given per predefined lung zone | at baseline and after 6 months of treatment
Total airway resistance for the segmented airways | at baseline and after 6 months of treatment

SECONDARY OUTCOMES:
BODE index | at baseline (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment (visit 8)
  The BODE index is a multidimensional index of disease severity . The index uses following parameters:
  * body mass index (BMI)
  * degree of airflow obstruction (Forced Expiratory Volume in 1 second (FEV1): % of predicted)
  * functional dyspnea (Modified Medical Reseach Council (MMRC) dyspnea scale)
  * exercise capacity (6 minute walk distance (6MWD) - m)
COPD assessment test | at screening (visit 1), at baseline (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment (visit 8)
  The COPD assessment measures the impact of COPD on a person's life.
Borg CR10 Scale | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
  The Borg CR10 Scale measures the present dyspnea.
Adverse events as a measure of safety | during the study patients will record record each day taken medication and any possible comments on the daily diary cards
  During the study patients will record record each day taken medication and any possible comments on the daily diary cards. Further more, patients are contacted at least once a month (either by phone or at a visit in the hospital).
Forced expiratory volume in 1 second (FEV1) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Forced Vital Capacity (FVC) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Peak Expiratory Flow (PEF) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Maximum expiratory flow rate at 50% of vital capacity (MEF50) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Maximal expiratory flow rate at 25% of vital capacity (MEF25) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Vital capacity (VC) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Inspiratory vital capacity (IVC) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Functional residual capacity (FRC) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Total Lung Capacity (TLC) | At screening, at baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Airway resistance (Raw) | At baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)
Specific airways conductance (SGaw) | At baseline both pre and post dose (visit 2), after 3 months of treatment (visit 5) and after 6 months of treatment both pre and post dose (visit 8)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD PhD, Principal Investigator — University Hospital of Antwerp
Locations (1):
- University Hospital of Antwerp, Edegem (Antwerp), Antwerp, Belgium